CLINICAL TRIAL: NCT02212275
Title: Initial Development of Cortical Metrics, an Objective, Physiologically-Based Outcome Measure, for Intervention Trials in Autism Spectrum Disorders (ASD)
Brief Title: Cortical Metrics in Intervention Trials With Autism Spectrum Disorders
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Duke University (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Pro00065239; 14-1141 (Other: UNC)
Record Dates: First submitted 2014-07-29; First posted 2014-08-08 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Autism Spectrum Disorders
Keywords: ASD; autism; typical development; sensory testing; the cortical metric
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dextromethorphan in ASD (Experimental): 8-12 years old: > 30 boys will be recruited who have a known or suspected diagnosis of ASD confirmed by DSM-5 checklist and the ADOS-2 at screening. They will have the cortical metric measured 20 min prior to receiving DXM and 2 hours after receiving a single age and weight appropriate dose of DXM. The outcome reported is the difference in the cortical metric after the DXM dose and before the DXM dose.
  Interventions: Drug: Dextromethophan
- Dextromethorphan in controls (Active Comparator): 30 typically developing boys 8-12 years old who have the cortical metric measured 20 min before receiving a single age and weight appropriate dose of DXM and 2 hours after the single dose of DXM. The reported value will be the difference between the cortical metric 2hrs after the single dose of DXM and the cortical metric 20 minutes prior to the single dose of DXM.
  Interventions: Drug: Dextromethophan

INTERVENTIONS:
Drug: Dextromethophan — A single age and weight appropriate dose of over the counter Delsym Cough Syrup containing only DXM as an active ingredient.
  Other Names: Delsym Cough Syrup

SUMMARY:
The investigators overarching aim is to obtain preliminary data to support a larger grant to validate a novel objective, physiologically-based outcome measure for clinical trials in autism spectrum disorders (ASDs) called the cortical metric. Absence of such an outcome measure has greatly hindered the development of treatments for core symptoms of ASD.

DETAILED DESCRIPTION:
The cortical metric is a single numeric measurement that is calculated using a multi-parametric mathematical approach from a series of measurements of the speed, intensity, diameter, and distance between two vibrations with which a person reacts to and can distinguish vibrations from small brushes that touch the top side of fingers on the left hand under multiple conditions designed to elicit cortical adaptation The cortical metric is based on the neurobiological principle that the nerves in the fingertips project to adjacent groups of neurons that work together to continuously optimize perceptions of touch under varying conditions. Such perceptual optimization reflects the shifting excitatory and inhibitory actions of individual neurons. We hypothesize that the brain's processing of vibration is similar to its processing of other kinds of information. We also hypothesize that in people with ASD adjacent groups of neurons work together less well to process information.

Specific Aim 1: Obtain evidence regarding the ability of the "cortical metric" to distinguish between 8-12 year-olds with typical development and with high functioning autism spectrum disorders (ASDs).

Hypothesis 1: The cortical metric of children with ASD will differ from that of age matched, typically developing children. This difference will be consistent with lower than normal local functional connectivity.

Specific Aim 2: Validate the test-retest reliability of the cortical metric by examining its stability of over an average of 3 weeks with no intervening interventions in both groups of children.

Hypothesis 2: Test-retest reliability will be highly correlated in both groups of children.

Specific Aim 3: Obtain preliminary proof of mechanism data that the cortical metric assesses the excitatory: inhibitory balance of intra-cortical connections by examining the effect of acute exposure to dextromethorphan (DXM), which transiently blocks one type of excitatory neurotransmission

Hypothesis 3: DXM will alter the cortical metric consistent with reduced adaptation.

The completion of these aims will be essential to design a larger federally funded trial to validate the cortical metric as an outcome measure in a more heterogeneous pediatric ASD sample. Specifically, we will aim to demonstrate that 1) the cortical metric differs between children with ASD and with normal development, 2) that the cortical metric has minimal variability over time in the absence of fno major changes in brain function, and 3) that the cortical metric changes in response to a specific, temporary reduction in excitatory stimulation caused by a single DXM dose.

A larger grant could focus on determining how sensitive and clinically relevant changes in the cortical metric are.

If we are not able to demonstrate the potential for the cortical metric to be changed by agents that reduce excitatory stimulation acutely or if the variability of the cortical metric over 3 weeks is too great, no further examination of the cortical metric as an outcome measure in ASD trials would be pursued. If there are not differences in the cortical metric of children with and without ASD, we would be less interested in further examining the cortical metric.

ELIGIBILITY:
Group 1 Typically Developing Youth: We will recruit 30 typically developing boys 8-12 years old to participate in a screening visit, and two tactile perception sessions (visit 1 and 2).

Inclusion Criteria:

* Healthy Male Boys ages 8-12
* Normal developmental milestones and school performance
* Primary caretaker is able to participate in study appointments as is indicated

Exclusion Criteria:

* Significant lifetime medical history including non-febrile seizures, neurological problems, psychiatric problems or learning disabilities
* Any sensory impairment (i.e. deafness or blindness)
* 1st or 2nd degree family members with a history of ASD
* 1st or 2nd degree family members with ADHD or other developmental problems
* Adverse reaction to dextromethorphan
* Inability to successfully complete and fully understand the reaction time subtest (cortical metrics)

Group 2 Youth with ASD: 8-12 years old: > 30 boys will be recruited who have a known or suspected diagnosis of ASD confirmed by DSM-5 checklist and the ADOS-2 at screening.

Inclusion Criteria:

* Male Boys ages 8-12 with ASD (confirmed by DSM-5 checklist and the ADOS-2)
* IQ's should be within the normal range (≥ 70) (by prior testing or Stanford Binet 5 at screening)
* Primary caretaker is able to participate in study appointments as is clinically indicated
* Ability of child to participate in all aspects of the protocol per investigator clinical judgment

Exclusion Criteria:

* New educational or behavioral intervention within 4 weeks of baseline
* History of non-febrile seizures, other neurological disorders, psychosis, bipolar disorder, or Tourette Syndrome.
* Any sensory impairment (i.e. deafness or blindness)
* Adverse reaction to dextromethorphan
* Inability to successfully complete and understand the reaction time subtest (cortical metrics)
* Changes in psychiatric medications within 4 weeks of baseline visit
* Taking epileptic medication (including but not limited to carbamazepine, phenobarbital, Depakote, lamictal, oxycarbazepine, topiramate)

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The difference in the Cortical Metric before and after acute exposure to dextromethorphan (DXM) | 2 hours after DXM exposure and 20 min before DXM
  At visit 2 the cortical metric will be measured 20 min prior to a single dose of DXM and 2hrs after the dose of DXM. . This addresses Specific Aim 3 of the trial. There are 3 primary outcomes all involving the cortical metric because the tool will not be useful to detect treatment changes unless all three outcomes demonstrate the desired response. Visit 2 occurs 3 weeks after baseline = time 0
Change in the cortical metric | 3 weeks
  The difference between the cortical metric measured 20 minutes before DXM treatment at visit 2, which occurs 3 weeks after the baseline = time 0 visit, and the cortical metric measured 3 weeks earlier at the baseline visit = time 0. We presume their will be no major changes in brain functioning over 3 weeks.
  This addresses Specific Aim 2 of the trial, regarding test retest stability. There are 3 primary outcomes all involving the cortical metric because the tool will not be useful to detect treatment changes unless all three outcomes demonstrate the desired response.
The Cortical Metric | Baseline = time 0
  The cortical metric will be measured at the baseline of the study = time 0. We will compare the mean cortical metric and the range of the cortical metric between the ASD and typically developing groups.
  This addresses Specific Aim 1 of the trial. There are 3 primary outcomes all involving the cortical metric because the tool will not be useful to detect treatment changes unless all three outcomes demonstrate the desired response. The goal of this aim is to replicate the findings of the John Hopkins University group that found differences in the cortical metric between groups of children 8-12 years old with ASD and with typical development.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC) Total Score | time 0 (baseline)
  The ABC focuses on problem behaviors in five subdomains: irritability, attention, repetitive behaviors, unusual speech, and social withdrawal and will be completed by subject's parent/guardian or caregiver.
  We will examine the correlation between the ABC Total score and the cortical metric.
Pervasive Developmental Disorders Behavior Inventory - Screening Version Score (PDDBI-SV) Social Deficit Score | Baseline = time 0
  The PDDBI-SV examines both adaptive and maladaptive behaviors related to autism. The adaptive items are reverse scored and then all items are summed to generate the social deficit score. It is not age specific. This questionnaire will be completed by subject's parent/guardian or caregiver. The correlation between the PDD-BI SV Social Deficit score and the cortical metric will be examined.
Social Responsiveness Scale, Version 2 Total Score (SRS) | Time 0 = Baseline
  This 65-item rating scale measures the severity of autism spectrum symptoms as they occur in natural social settings (Constantino, Davis et al. 2003). Completed by a parent or teacher in just 15 to 20 minutes, the SRS provides a clear picture of a child's social impairments, assessing social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance, and autistic preoccupations and traits. It is appropriate for use with children from 4 to 18 years of age. The SRS measures impairment on a quantitative scale across a wide range of severity--which is consistent with recent research indicating that autism is best conceptualized as a spectrum condition rather than an all-or-nothing diagnosis. This will be completed by the subject's parent/guardian or caregiver.
  The correlation between the SRS Total score and the cortical metric will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke Center for Autism and Brain Development, Durham, North Carolina